CLINICAL TRIAL: NCT01506531
Title: Bedside Silo Versus Attempted Operative Closure for Gastroschisis
Brief Title: Silo Versus Primary Closure for Gastroschisis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Shawn St. Peter, Associate Professor, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11 09-156
Record Dates: First submitted 2012-01-02; First posted 2012-01-10 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Gastroschisis
Keywords: gastroschisis; silo; primary closure
MeSH Terms: conditions — Gastroschisis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- primary closure of gastroschisis (Active Comparator): Attempt primary skin closure of gastroschisis shortly after birth
  Interventions: Procedure: Primary closure of gastroschisis
- silo for gastroschisis (Active Comparator): Surgical placement of silo over gastroschisis shortly after birth
  Interventions: Procedure: silo for gastroschisis

INTERVENTIONS:
Procedure: silo for gastroschisis — silo placed around abdominal contents in gastroschisis patients
  Arms: silo for gastroschisis
Procedure: Primary closure of gastroschisis — Primary closure of gastroschisis, if possible
  Arms: primary closure of gastroschisis

SUMMARY:
The objective of this study is to scientifically evaluate two different closure strategies for gastroschisis to determine if there is a difference in the two approaches.

DETAILED DESCRIPTION:
The hypothesis is that there is no difference between bedside silo placement and operative closure in return of bowel function, ventilator dependence, or length of stay.

The primary outcome variable between the two techniques will be length of hospitalization. The likely variables will be length of time to meet discharge criteria, length of hospitalization, time to full feedings, time on mechanical ventilation and total hospital charges.

ELIGIBILITY:
Inclusion Criteria:

* Infants with gastroschisis

Exclusion Criteria:

* Born prior to 34 weeks estimated gestational age
* Another congenital anomaly influencing the respiratory status, gastrointestinal status, or the length of hospitalization and recovery.
* Inability to get parental permission before treatment.

Ages: 5 Minutes to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Length of hospitalization | 1-6 weeks
  The length of time required for meeting discharge criteria

CONTACTS AND LOCATIONS:
Overall Officials: Shawn D St. Peter, MD, Principal Investigator — Children's Mercy Hospital and Clinics
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No